CLINICAL TRIAL: NCT03678363
Title: Effect of Tai Chi Protocol on Total Physical Activity in Patients With Rheumatoid Arthritis, in Comparison With a Control Group Without Tai Chi.
Brief Title: Tai Chi in Rheumatoid Arthritis (TaiChiRA)
Acronym: TaiChiRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHU-400; 2017-A03294-49 (Other: 2017-A03294-49)
Record Dates: First submitted 2018-07-12; First posted 2018-09-19 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Tai chi chuan; Physical Activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Tai Ji

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group A (Experimental): 2 tai chi session per week during 4 month (M0 to M4)
  Interventions: Other: Tai chi chuan
- Control group B (Placebo Comparator): 2 tai chi session per week during 2 month (M2 to M4)
  Interventions: Other: Tai chi chuan

INTERVENTIONS:
Other: Tai chi chuan — Tai chi sessions will consist of repetition of simple and basic movements focusing mainly on breating, relaxation and body diagram. This Chinese martial art also includes coordination exercises of body parts (legs, arms, pelvis and spine), looseness and limbering up of joints and muscles.

SUMMARY:
The investigator's hypothesis is that tai chi sessions would increase physical activity of patients with Rheumatoid Arthritis. The main objective is to study the effect of tai chi sessions (16 vs.0) on total physical activity of Rheumatoid Arthritis patients, compared to a control group without tai chi.

DETAILED DESCRIPTION:
Detail protocol:

Selection and inclusion of patients will be done by principal investigator of Rheumatology Department. After verification of inclusion and non-inclusion criteria by principal investigator and signature of consent, patients will be randomized by 1: 1 randomization (centralized randomization by statistician into 2 groups at Month 0). They will participate in sessions in a deferred manner due to two per week for each group:

* Interventional "A" group: 32 sessions (on average 2/week) performed from Month 0 to Month 4 in 15 patients.
* Control "B" group: 16 sessions (on average 2/week) performed from Month 2 to Month 4 in 15 patients.

Patients of "B" group will be not performing sessions with "A" group patients. Sessions lasting about 45 minutes will be proposed from Monday to Friday in a room planned from this activity within the CHU. Exercises will be adapted and personalized according to each one. Evaluations will be carried out for group 1 (interventional) before the first session of tai chi at Month 0, before the session at Month 2 and at the end of the protocol at Month 4. The same evaluations will be carried out for group B (control) at Month 0, before first session of tai chi at Month 2 and at the end of the protocol.

Assessment of pain and stress will be done before and after each session. Final assessment will be done at 4 months after randomization. Fitness assessment and tai chi sessions will be conducted by APA student. Clinical examination of patient, installation and removal of cardio frequency meter will be performed by nurse. Data entry will be done by Clinical Research Associate of the Rheumatology Department. Statistical analysis will be carried out by biostatistician affiliated to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old with RA (ACR/EULAR criteria) in remission (CDAI ≤2.8) or with low disease activity (CDAI ≤10).
* Patient able to walk without help
* Patient able to complete a questionnaire
* Patient giving informed consent.
* Patient covered by social security

Exclusion Criteria:

* Patient with disorder of higher mental function or psychiatric disorders.
* Patient who has previously contribute to a tai chi program.
* Patient with an absolute contraindication to physical activity.
* Protected populations: pregnant women, breastfeeding women, tutorship, trusteeship, deprived of liberty, safeguard of justice.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-31 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in total physical activity time expressed in min/ day between M0 and M2 measured by eMouve smartphone application | At Month 0 before the first session of tai chi and Month 2 after 16 sessions of tai chi (intervention group), measured at Month 0 and Month 2 (control group without tai chi).
  Android application allows to estimate in usual conditions of life the energy expenditure and time spent in three intensities of physical activities: light, moderate and vigorous, as well as the time spent in sedentary behaviors. Android smartphone with application eMouve will be entrusted to patients to collect information from their physical activity (PA) for 4 days (2 days of the week and 2 days of weekend).
Change in total physical activity time expressed in MET.min/week between M0 and M2 measured by Global physical activity questionnaire (GPAQ Questionnaire (Global Physical Activity Questionnaire) | At Month 0 before the first session of tai chi and Month 2 after 16 sessions of tai chi (intervention group), measured at Month 0 and Month 2 (control group without tai chi).
  Modified Global Physical Activity Questionnaire provides a longitudinal assessment of a typical week for physical activity and sedentary behaviors. It covers three areas of activities: work activity, utilitarian travel, leisure activities and home-based activities. This questionnaire provides information on time spent on different activities in each of three areas mentioned above. A specific energy expenditure is associated with each PA, which makes it possible to estimate the overall energy expenditure of the patients. It also provides information on sedentary time.

SECONDARY OUTCOMES:
Disease activity, evaluated by CDAI score (Clinical Disease Activity Index) at M0, at M2 after 16 sessions and at M4 after 32 sessions (interventional group) and evaluated at M0, M2 and M4 after 16 sessions (control group). | at M0, M2 and M4 after 16 sessions
  CDAI score (Clinical Disease Activity Index) corresponds to the algebraic sum of the number of painful (N=28) and swollen (N=28) joints, of disease activity judged by patient on analogical visual scale (AVS) from 0 to 10 cm and disease activity on AVS from 0 to 10cm evaluated by the physician. Remission is defined by a score ≤ 2.8 and low activity by a score ≤ 10.
Sedentary time expressed in ME.min/week measured by modified Global Physical Activity Questionnaire. | At Month 0, Month 2 after 16 sessions and at Month 4 after 32 sessions (interventional group) and measured at Month 0, Month 2 and Month 4 after 16 sessions (control group).
  Modified Global Physical Activity Questionnaire provides a longitudinal assessment of a typical week for physical activity and sedentary behaviors. It covers three areas of activities: work activity, utilitarian travel, leisure activities and home-based activities. This questionnaire provides information on time spent on different activities in each of three areas mentioned above. A specific energy expenditure is associated with each PA, which makes it possible to estimate the overall energy expenditure of the patients. It also provides information on sedentary time.
Physical activity time of light intensity, moderate intensity, high intensity measured by the modified GPAQ expressed in ME.minute/week | At Month 0, at Month 2 after 16 sessions and at Month 4 after 32 sessions (interventional group) and measured at Month 0, Month 2 and Month 4 after sessions (control group).
  Modified Global Physical Activity Questionnaire provides a longitudinal assessment of a typical physical activity and sedentary behaviors. It covers three areas of activity: work activity, utilitarian travel, leisure activities and home-based activities. This questionnaire provides information on time spent on different activities in each of three areas mentioned above. A specific energy expenditure is associated with each PA which allows to estimate the overall energy expenditure of the patients. It also provides information on sedentary time.
Schober test | At Month 0, at Month 2 after 16 sessions and at Month 4 after 32 sessions (group interventional) and measured at Month 0, Month 2 and Month 4 after 16 sessions (control group).
  Schober test consists of evaluating flexion amplitude of lumbar spine: two marks are made at L5 vertebra and 10cm above this lumbar vertebra, in a standing patient. Patient is then asked to lean forward and measure the increase in gap between two marks previously practiced. A gap of less than 3cm is considered pathological, the expected normal is +5cm.
The single leg stance test | At Month 0, at Month 2 after 16 sessions and at Month 4 after 32 sessions (group interventional) and measured at Month 0, Month 2 and Month 4 after 16 sessions (control group).
  Subject must stand unassited on one leg and is timed in seconds from the time one foot is flexed off the floor to the time when it touches the ground or the standing leg or an arm leaves the hip. Goal is to maintain a balance as long as possible. Test is performed on each leg with eyes open and eyes closed.
6 minutes walk test | At Month 0, at Month 2 after 16 sessions and at Month 4 after 32 sessions (group interventional) and measured at Month 0, Month 2 and Month 4 after 16 sessions (control group).
  The 6 minutes walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Handgrip strengh test | At Month 0, at Month 2 after 16 sessions and at Month 4 after 32 sessions (group interventional) and measured at Month 0, Month 2 and Month 4 after 16 sessions (control group).
  Muscular strength of both hands will be measured by dynamometry. Dynamometer electronics interpret voltage to display it as a unit of force. Best of three tries on each side is retained and scored (one value for each slide).
Sit-to-stand test | At Month 0, at Month 2 after 16 sessions and at Month 4 after 32 sessions (group interventional) and measured at Month 0, Month 2 and Month 4 after 16 sessions (control group).
  Muscle strength of lower limbs will be measured by sit-to-stand test. Participant sits in middle of a chair, his back straight, his feet flat on the floor. Arms are crossed and hands resting on the chest. At the signal, participant gets up completely before sitting down in the initial position. He is invited to realize the maximum of lifts during 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Martin SOUBRIER, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Cleland CL, Hunter RF, Kee F, Cupples ME, Sallis JF, Tully MA. Validity of the global physical activity questionnaire (GPAQ) in assessing levels and change in moderate-vigorous physical activity and sedentary behaviour. BMC Public Health. 2014 Dec 10;14:1255. doi: 10.1186/1471-2458-14-1255. PMID 25492375
- [Background] Ekelund U, Steene-Johannessen J, Brown WJ, Fagerland MW, Owen N, Powell KE, Bauman A, Lee IM; Lancet Physical Activity Series 2 Executive Committe; Lancet Sedentary Behaviour Working Group. Does physical activity attenuate, or even eliminate, the detrimental association of sitting time with mortality? A harmonised meta-analysis of data from more than 1 million men and women. Lancet. 2016 Sep 24;388(10051):1302-10. doi: 10.1016/S0140-6736(16)30370-1. Epub 2016 Jul 28. PMID 27475271
- [Background] Gossec L, Paternotte S, Aanerud GJ, Balanescu A, Boumpas DT, Carmona L, de Wit M, Dijkmans BA, Dougados M, Englbrecht M, Gogus F, Heiberg T, Hernandez C, Kirwan JR, Mola EM, Cerinic MM, Otsa K, Schett G, Scholte-Voshaar M, Sokka T, von Krause G, Wells GA, Kvien TK. Finalisation and validation of the rheumatoid arthritis impact of disease score, a patient-derived composite measure of impact of rheumatoid arthritis: a EULAR initiative. Ann Rheum Dis. 2011 Jun;70(6):935-42. doi: 10.1136/ard.2010.142901. PMID 21540201
- [Background] Guidoux R, Duclos M, Fleury G, Lacomme P, Lamaudiere N, Manenq PH, Paris L, Ren L, Rousset S. A smartphone-driven methodology for estimating physical activities and energy expenditure in free living conditions. J Biomed Inform. 2014 Dec;52:271-8. doi: 10.1016/j.jbi.2014.07.009. Epub 2014 Jul 15. PMID 25048352
- [Background] Guidoux R, Duclos M, Fleury G, Lacomme P, Lamaudiere N, Saboul D, Ren L, Rousset S. The eMouveRecherche application competes with research devices to evaluate energy expenditure, physical activity and still time in free-living conditions. J Biomed Inform. 2017 May;69:128-134. doi: 10.1016/j.jbi.2017.04.005. Epub 2017 Apr 9. PMID 28400313
- [Background] Jones SD, Porter J, Garrett SL, Kennedy LG, Whitelock H, Calin A. A new scoring system for the Bath Ankylosing Spondylitis Metrology Index (BASMI). J Rheumatol. 1995 Aug;22(8):1609. No abstract available. PMID 7473496
- [Background] Uhlig T. Tai Chi and yoga as complementary therapies in rheumatologic conditions. Best Pract Res Clin Rheumatol. 2012 Jun;26(3):387-98. doi: 10.1016/j.berh.2012.05.006. PMID 22867933
- [Background] Veldhuijzen van Zanten JJ, Rouse PC, Hale ED, Ntoumanis N, Metsios GS, Duda JL, Kitas GD. Perceived Barriers, Facilitators and Benefits for Regular Physical Activity and Exercise in Patients with Rheumatoid Arthritis: A Review of the Literature. Sports Med. 2015 Oct;45(10):1401-12. doi: 10.1007/s40279-015-0363-2. PMID 26219268
- [Background] Waite-Jones JM, Hale CA, Lee HY. Psychosocial effects of Tai Chi exercise on people with rheumatoid arthritis. J Clin Nurs. 2013 Nov;22(21-22):3053-61. doi: 10.1111/jocn.12327. Epub 2013 Sep 13. PMID 24033836
- [Background] Wang C. Role of Tai Chi in the treatment of rheumatologic diseases. Curr Rheumatol Rep. 2012 Dec;14(6):598-603. doi: 10.1007/s11926-012-0294-y. PMID 23055009
- [Background] Wang C. Tai Chi improves pain and functional status in adults with rheumatoid arthritis: results of a pilot single-blinded randomized controlled trial. Med Sport Sci. 2008;52:218-229. doi: 10.1159/000134302. PMID 18487901